CLINICAL TRIAL: NCT03790163
Title: The Influence of Different Degrees of Levobupivacaine Temperature on Spinal Anesthesia in Orthopedic Surgeries: Prospective Randomized Study
Brief Title: The Effect of Different Degree of Temperature on Levobupivacaine Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Abdelraouf Elsharkawy, Lecturer of anesthesia and surgical intensive care, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MFM.IRB,R/18.11.340
Record Dates: First submitted 2018-12-24; First posted 2018-12-31 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Spinal Anesthetic Toxicity
Keywords: levobupivacaine,spinal anesthesia ,temperature
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double(participant ,care provider)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- levobupivacaine at ( 23˚C) (Placebo Comparator): Levobupivacine hydrochloride at ( 23˚C) will be received 3.5 ml levobupivacaine at the operating room temperature 23˚C will be administered
  Interventions: Drug: Levobupivacaine
- Warm levobupivacaine at (30˚C) (Active Comparator): Drug:Warm levobupivacaine hydrochlorid (3.5 ml) will be warmed at (30˚C) for 24 hours. The empty syringes and needles ,in their packaging, will be held at the same temperature before the spinal anesthesia
  Interventions: Drug: Levobupivacaine
- Warm levobupivacaine at (37˚C) (Active Comparator): Drug:Warm levobupivacaine hydrochlorid (3.5 ml) will be warmed at (37˚C) for 24 hours. The empty syringes and needles ,in their packaging, will be held at the same temperature before the spinal anesthesia
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Drug: levobupivacaine at room temperature ( 23˚C) and second group levobupivacaine warmed to the (30˚C) while the third group levobupivacaine warmed to the body temperature (37˚C)
  Other Names: Chirocaine

SUMMARY:
This study will be conducted to evaluate the effect of different temperature on the spinal anesthesia characteristics and incidence of complications

DETAILED DESCRIPTION:
Regional anesthesia techniques are also superior to systemic opioids agents with regard the analgesic profile and adverse effects .Spinal anesthesia is the most commonly used technique due to its unmatchable reliability,simplicity and cost-effectiveness. It provides a fast and effective onset of sensory and motor block, excellent muscle relaxation and prolonged postoperative analgesia .

Bupivacaine is commonly used local anesthetics because of its long duration of action and combined motor and sensory blockade. However, it has many drawbacks .It has a high propensity to cause hypotension and bradycardia. There is also cardiac toxicity.Levobupivacaine is an attractive alternative to bupivacaine because of the lower affinity for cardiac sodium channels and reducing the risk of cardiac toxicity.Moreover ,the isobaric levobupivacaine had more stability in cerebrospinal fluid and thus lead to more predictable drug spread, decreasing the incidence of hypotension and bradycardia. But its main disadvantage is the delayed onset .

A number of strategies have been used to hasten the onset of local anesthesia .The addition of fentanyl mixtures of local anesthetics and alkalization of the local anesthetics all shorten the onset time of sensory block. Recently the warming of the anesthetic agents (namely, lidocaine and bupivacaine) to 37° C hastens the sensory block in various surgical settings .

Up till now there is no study suggestive of any appropriate degree of temperature as adjuvant .Hence the present study will be conducted to evaluate the effect of different temperature on spinal anesthesia characteristics and the incidence its complication

ELIGIBILITY:
Inclusion Criteria:

* ASA-I or II

Exclusion Criteria:

* patient refusal; Any known hypersensitivity or contraindication to levobupivacaine pregnancy bleeding disorders local skin infections. Sepsis at the site of injection Coagulation abnormality Psychiatric disorders

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-15 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Time to onset of sensory block | For 10 minutes following the spinal anesthesia
  Defined as the time interval between the end of spinal anesthesia injection and the loss of sensation to pin prick (sensory score=1)

SECONDARY OUTCOMES:
Time to the onset of motor block | For 10 minutes following the injection of spinal anesthesia
  Defined as the time interval between the end of spinal anesthesia and (motor score=1) within both lower limbs
Duration of sensory block | For 24 hours after the spinal anesthesia
  Defined as the interval between the end of spinal anesthesia and complete end of sensory block (sensory score=2)
Duration of motor block | For 24 hours after the spinal anesthesia
  Defined as the interval between the end of spinal anesthesia and complete recovery of normal motor function (score=0)
Post spinal shivering | for 24 hours after spinal anesthesia
  Post spinal shivering will be graded using a scale ( score 0=no shivering ,score 1= no visible muscle activity ,but one or more of piloerection, score 2=muscular activity in only one muscle group,score 3=moderate muscular activity in more than one muscle group but not generalized shaking ,score 4=violent muscular activity that involves entire body )

CONTACTS AND LOCATIONS:
Overall Officials: Reem El sharkawy, Principal Investigator — lecturer of anesthesia and surgical intensive care ,faculty of medicine
Locations (1):
- Adham Elgeidi, Al Mansurah, Dakahliah, Egypt